CLINICAL TRIAL: NCT06612034
Title: Evaluating the Worldwide Landscape of Prostate Cancer Management
Brief Title: Prostate Cancer Care Disparity Analysis Project (ProGAP)
Status: Recruiting | Type: Observational
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Yüksel Ürün, Professor doctor, Ankara University
Other Study IDs: ANKARA-UNIVERSITY-YURUN-01
Record Dates: First submitted 2024-09-21; First posted 2024-09-25 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2024-09

CONDITIONS: Prostate CA
Keywords: prostate cancer; Human Development Index; survey; access to medicine; multidisciplinary care
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Healthcare professionals for prostate cancer: Healthcare professionals actively engaged in prostate cancer treatment, including urologists, uro-oncologists, medical oncologists, and radiation oncologists
  Interventions: Other: No Intervention: Observational Cohort

INTERVENTIONS:
Other: No Intervention: Observational Cohort — No Intervention: Observational Cohort

SUMMARY:
This international cross-sectional study seeks to evaluate global disparities in prostate cancer management by conducting a thorough comparison of key elements across countries categorized as low-income, lower-middle-income, upper-middle-income, and high-income.

The primary question it addresses is: Are the standards of care for prostate cancer uniformly applied across different geographic regions worldwide? To achieve this, we will recruit physicians specializing in the diagnosis and treatment of prostate cancer from a diverse array of countries within these income classifications. Participants will complete a 17-question online survey.

DETAILED DESCRIPTION:
Prostate cancer stands as one of the most common cancers among men worldwide, with outcomes and care quality significantly varying due to a multitude of factors including geographic location, healthcare infrastructure, socioeconomic status, and clinical practices. The ProGAP project is conceived to delve into these variations, providing a detailed examination of the global landscape of prostate cancer care.

Objectives:

1. To systematically gather and analyze data on current diagnostic methods, treatment modalities, and management practices for prostate cancer from a wide range of countries and healthcare settings.
2. To identify and quantify disparities in access to and availability of standard care, novel treatments, and supportive services for patients with prostate cancer.
3. To evaluate the adherence levels to both international and national guidelines in prostate cancer treatment across diverse healthcare systems.

Methods:

The ProGAP survey will be distributed internationally to healthcare professionals, including urologists, uro-oncologists, medical oncologists, and radiation oncologists, who are actively involved in prostate cancer care. The survey will comprehensively cover demographic details, clinical practice environment, patient demographics and stages managed, guideline adherence, availability and use of diagnostic and treatment options, and multidisciplinary care approaches. A survey and a consent form will be sent to study participants in addition to written information about the study. Completing surveys will take 10-12 minutes. Participants will complete a 17-question online survey. The first part of the form includes questions about demographics and hospital characteristics. The second part contains questions about prostate cancer diagnosis, treatment, and management practices. Participation in this study is entirely voluntary and anonymous. Neither sensitive personal data nor contact information will be collected during the research. This research does not receive any specific grant from funding agencies in the public, commercial, or not-for-profit sectors, and the investigators declare that they do not have any conflict of interest with the work.

Data Analysis Plan:

Statistical analyses will employ both descriptive and inferential statistics to interpret the survey data. Comparative analyses will be conducted to uncover disparities across different regions and healthcare settings. Advanced statistical methods, such as regression analysis, may be utilized to explore factors associated with variations in care practices and outcomes.

Expected Impact:

By elucidating the disparities in prostate cancer care worldwide, ProGAP aims to stimulate policy changes, guide improvements in clinical practice, and foster international collaborations to enhance the quality of care and outcomes for patients with prostate cancer globally. Insights gained from this project are anticipated to inform stakeholders, including healthcare providers, policymakers, and patient advocacy groups, about critical areas for intervention and improvement.

ELIGIBILITY:
Inclusion Criteria:

Urologists, Uro-oncologists, Medical oncologists, Radiation oncologists

Exclusion Criteria:

Non-clinical healthcare professionals Healthcare professionals not directly involved in the care of prostate cancer patients, Healthcare professionals with missing or incorrect email addresses

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthcare professionals actively treating prostate cancer patients-such as urologists, uro-oncologists, medical oncologists, and radiation oncologists-who specialize in the diagnosis and treatment of prostate cancer, representing a diverse range of countries categorized as low-income, lower-middle-income, upper-middle-income, and high-income
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Characterization of global disparities in prostate cancer diagnosis, treatment, and management practices | One month
  Comparative analyses will be conducted using survey data to reveal disparities between different regions and healthcare settings. The findings will be presented as percentages of respondents, with territorial and institutional differences thoroughly evaluated. Participants will be categorized into three groups based on the World Bank's income classification: low and lower-middle, upper-middle, and high-income countries. Descriptive statistics will be employed to compare demographic characteristics and clinical practices. For categorical data analysis, the Pearson Chi-Square or Fisher's Exact test will be utilized, while ANOVA tests will be applied to independent variables. A p-value of less than 0.05 will be considered statistically significant.

SECONDARY OUTCOMES:
Assessment of access to care, encompassing advanced diagnostic tools, treatment modalities, and patient support services; analysis of adherence to guidelines and its effect on treatment outcomes | One month
  Identifying the percentage of healthcare professionals across various geographic regions who have access to diagnostic and treatment methods that align with established guidelines, and evaluating the impact of these methods on treatment outcomes. The findings will be presented as percentages of respondents, with territorial and institutional differences thoroughly examined.

CONTACTS AND LOCATIONS:
Overall Officials: Yüksel Ürün, Study Director — Ankara University; Deborah Mukherji, Study Director — Clemenceau Medical Center Hospital Dubai; Mohammed Shahait, Study Director — Al Zahra Hospital Dubai; Luis Castelo Branco, Study Director — IOSI Oncologist Institute of Southern Switzerland
Locations (1):
- Ankara University Faculty of Medicine, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The data that support the findings of this study are available from the study director upon reasonable request.